CLINICAL TRIAL: NCT02928471
Title: Multi-parametric Imaging of the Knee in Obese Patients With Knee Osteoarthritis Following a Significant Weight Loss, Investigating the Impact on Inflammation (A Substudy to "Effect of Liraglutide on Body Weight and Pain in Overweight or Obese Patients With Knee Osteoarthritis: A Randomised, Double Blind, Placebo-controlled, Parallel Group, Single-centre Trial" (NCT02905864)
Brief Title: Multi-parametric Imaging of the Knee in Obese Patients With Knee Osteoarthritis; Weight Loss
Acronym: IM-LOSEIT-I
Status: Completed | Type: Observational
Sponsor: Henrik Gudbergsen (Other)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Organization: Parker Research Institute (Other)
Other Study IDs: 137.03
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis; Obesity
Keywords: Liraglutide; Liraglutide 3 mg; Osteoarthritis; Obesity; Magnetic resonance imaging; Computed tomography; Dynamic contrast enhanced MRI
MeSH Terms: conditions — Osteoarthritis; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intensive dietary intervention: Supervised dietary weight loss program lasting 8 weeks.
  Interventions: Dietary Supplement: Intensive dietary intervention

INTERVENTIONS:
Dietary Supplement: Intensive dietary intervention — Participants receive a hypo-caloric formula diet containing 800 to 1,000 kcal/day. The formula diet consists of ready-to-use meal bars and powders to mix with water to make shakes, soups, or porridge. The weight loss programme consists of an 8-week period with full meal replacement by a standard liquid energy intake protocol. To facilitate compliance with the programme, participants will be scheduled for weekly facility-based group sessions with 6-8 participants led by a dietician. The recommendations for daily nutrient intake will be met.

SUMMARY:
This is a substudy to a randomised trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis (NCT02905864). In the parent trial, patients will be subjected to an 8-week diet intervention phase including a low-calorie diet and dietetic counseling, after which. Patients will be randomised to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

This substudy aims to investigate any changes in MRI associated with the initial 8-week weight loss intervention, and the value of CT scans in predicting the effect of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Same as parent trial (NCT02905864)

Further Exclusion Criteria

* Same as parent trial (NCT02905864)
* Usual exclusion criteria for MRI (i.e. pacemakers etc.)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants eligible for parent trial (NCT02905864), i.e. overweight/obese individuals with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in the degree of inflammation in the knee-joint (DCE-MRI) | Week -8 to 0
  Change will be assessed via a dynamic contrast enhanced MRI evaluation of corpus hoffa (Ballegaard C et al. and Riis RG et al.)

SECONDARY OUTCOMES:
Change in the degree of inflammation in the knee-joint (CE-MRI) | Week -8 to 0
  Change will be assessed via a static contrast enhanced MRI evaluation of the level of synovitis in the knee-joint (11 sites scored 0-2, ad modum Guermazi et al.)
Change in the degree of inflammation in the knee-joint (MRI) | Week -8 to 0
  Change will be assessed via a conventional MRI evaluation of the level of synovitis and effusion (combined) in the knee-joint (MOAKS)
Change in cartilage composition | Week -8 to 0
  Change will be assessed via T2-maps of cartilage in the weight-bearing parts of the knee-joint (ROI)
Change in bone marrow lesions (BML) | Week -8 to 0
  Change will be assessed via the MRI knee scoring system MOAKS; BML sum-score
Prediction of clinical symptoms (KOOS pain) by the level of crystal deposition on dual-energy CT at week 0 | Week 0
  Crystal deposition will be evaluated via dual-energy CT

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute and Department of Radiology at Bispebjerg and Frederiksberg Hospital, Frederiksberg, Capital Region, Denmark